CLINICAL TRIAL: NCT05150535
Title: A Prospective Study of One Week Accelerated Hypo-fractionation Adjuvant Radiotherapy in High-risk Breast Cancer Patients
Brief Title: One Week Adjuvant Radiotherapy for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Elmahdy, Assistant lecturer of clinical oncology sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21_10_18
Record Dates: First submitted 2021-11-03; First posted 2021-12-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionation control arm (Active Comparator): Patients who will receive 40 Gy in 15 fractions to the entire breast or chest wall over three weeks and have had breast conservation surgery (BCS) or oncoplastic breast surgery(OBS) will receive an additional boost to the tumour site if and will receive sequential dose 12GY\4 fractions or SIB 8GY 15 fractions. The supraclavicular fossa will be treated in patients with node-positive disease or those who had received neoadjuvant chemotherapy . The IMLN will be irradiated in N2and N3 at first presentation.
  Interventions: Radiation: Hypofractionation Radiotherapy.
- . Ultrahypofractionation experimental arm (Experimental): Patients who will receive 26 Gy in 5 fractions to the entire breast and or chest wall for one week only. The volume of this arm will be the same as the volume of the control arm as regard axillary nodes, supraclavicular and IMLN. Patients who have had breast conservation or oncoplastic breast surgery(OBS) will be given a boost. If a boost is given, SIB of 6 Gy in 5 fractions will be used (or a sequential boost of 12GY\4 fractions).
  Interventions: Radiation: Ultra-hypofractionation radiotherapy

INTERVENTIONS:
Radiation: Hypofractionation Radiotherapy. — Patients will receive 40 Gy in 15 fractions to the entire breast and or chest wall over the course of 3 weeks.
  Other Names: 3 weeks radiotherapy.
  Arms: Hypofractionation control arm
Radiation: Ultra-hypofractionation radiotherapy — Patients will receive 26 Gy in 5 fractions to the entire breast and or chest wall over the course of one week.
  Other Names: 1 week accelerated hypo-fractionation radiotherapy
  Arms: . Ultrahypofractionation experimental arm

SUMMARY:
* Cancer is the second leading cause of death after cerebrovascular strokes and is a significant obstacle to each nation's future growth.
* Worldwide, Breast cancer is the most common cancer in women and the 5th leading cause of cancer related deaths that comes after lung cancer, colorectal cancer, liver cancer and gastric cancer.
* More than half of all breast cancer cases in the world occur in developing countries. Egypt has a high mortality rate from breast cancer, with a rate of 21.3 per 100,000 cases. Breast cancer is diagnosed at an advanced stage in 60 to 70% of cases in Egypt. The median age at diagnosis in Egypt is 48.5 years, which seems to be a decade younger than in Europe and North America.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 45 years of age or older who have had Oncoplastic Breast Surgery (OBS) or total mastectomy with adequate axillary clearance and a negative margin.
* Breast carcinomas that is invasive (TXN1-3M0, T0N2-3 M0, T1N2-3M0, T2N2-3M0, T3N0-3M0, T4N0-3M0) whatever type of tumors biology.
* All patients with locally advanced breast cancer who received neoadjuvant chemotherapy and underwent either oncoplastic breast surgery or modified radical mastectomy

Exclusion Criteria:

* Metastatic breast cancer at the time of diagnosis proved clinically or radiologically.
* Postoperative positive margin.
* Carcinomas in situ.
* Mesenchymal breast lesions.
* Locoregional recurrent breast cancer.
* Synchronous bilateral breast cancer.
* very early breast cancer (T1-2N0M0,T1N1M0).

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female adult patients with breast
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months
  Rate of acute grade 2 toxicity or higher from the treatment till 3 months (NCI_CTCAE).
  Each patient will be assesed weekly during radiotherapy and monthly for 3 months post radiotherapy.
Chronic toxicity | 6 months post treatment up to 2 years
  Rate of chronic toxicity grade 2 or higher ( NCI_CTCAE) from 6 months after radiotherapy up to 2 years.
  Each patient will be assessed before treatment and at 6,12 and 24 months from treatment.
Local recurrence | Up to 2 years
  Rate of ipsilateral locoregional tumor recurrence proved by imaging and biopsy.
Patient compliance | From the starting point of treatment till the end of treatment ( 3 weeks in control arm and 1 week in experimental arm
  Compliance to treatment (number of interrupted days of radiotherapy.

SECONDARY OUTCOMES:
Overall survival | From time of diagnosis up to 2 years post radiotherapy
  Overall survival (Number of the surviving patients for 2 years in each arm of the study)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gany F, Ayash C, Raad N, Wu M, Roberts-Eversley N, Mahmoud H, Fouad Y, Fahmy Y, Asar H, Salama A, El-Shinawi M. Financial and food security challenges of Egyptian women undergoing breast cancer treatment. Support Care Cancer. 2020 Dec;28(12):5787-5794. doi: 10.1007/s00520-020-05426-9. Epub 2020 Mar 27. PMID 32221669
- [Background] Momenimovahed Z, Salehiniya H. Epidemiological characteristics of and risk factors for breast cancer in the world. Breast Cancer (Dove Med Press). 2019 Apr 10;11:151-164. doi: 10.2147/BCTT.S176070. eCollection 2019. PMID 31040712
- [Background] Stapleton SM, Oseni TO, Bababekov YJ, Hung YC, Chang DC. Race/Ethnicity and Age Distribution of Breast Cancer Diagnosis in the United States. JAMA Surg. 2018 Jun 1;153(6):594-595. doi: 10.1001/jamasurg.2018.0035. PMID 29516087